CLINICAL TRIAL: NCT02239172
Title: A Phase 1 Study of the Safety and Immunogenicity of Plant-Derived Recombinant Protective Antigen (rPA) Anthrax Vaccine in Healthy Adults
Brief Title: PA83-FhCMB Plant-Derived Recombinant Protective Antigen (rPA) Anthrax Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fraunhofer, Center for Molecular Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: FhCMB rPA83-001
Record Dates: First submitted 2014-08-13; First posted 2014-09-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Anthrax
MeSH Terms: conditions — Anthrax

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 12.5 µg + Alhydrogel (Experimental): vaccine
  Interventions: Biological: PA83-FhCMB
- 25 µg + Alhydrogel (Experimental): vaccine
  Interventions: Biological: PA83-FhCMB
- 50 µg + Alhydrogel (Experimental): vaccine
  Interventions: Biological: PA83-FhCMB
- 100 µg + Alhydrogel (Experimental): vaccine
  Interventions: Biological: PA83-FhCMB

INTERVENTIONS:
Biological: PA83-FhCMB

SUMMARY:
The purposes of this study is to evaluate and compare the safety, reactogenicity, and tolerability of the PA83-FhCMB vaccine candidate delivered at 4 dose levels with Alhydrogel

ELIGIBILITY:
Inclusion Criteria:

* Citizen or permanent resident of the US
* Male or female aged 18 to 49 years inclusive
* Able to give written informed consent
* Healthy, as determined by medical history, physical examination, vital signs, and clinical safety laboratory examinations at baseline
* Females should fulfill one of the following criteria:

  1. At least one year post-menopausal
  2. Surgically sterile
  3. Willing to use a medically approved form of contraception (eg, oral, implantable, transdermal, or injectable hormonal contraceptive; intrauterine device; barrier protection to include female condom, diaphragm, cervical cap, or male condoms in conjunction with spermicide) for 30 days prior to first vaccination and through the end of the study
  4. Willing to abstain from sexual intercourse for 30 days prior to first vaccination and through the end of the study
* Women of childbearing potential must have a negative urine pregnancy test within 24 hours preceding receipt of each dose
* Comprehension of the study requirements
* Expressed availability for the required study period
* Ability to attend scheduled visits and to be contacted by telephone throughout the follow-up period

Exclusion Criteria:

* History of anthrax disease or receipt of anthrax vaccine
* Presence of significant uncontrolled medical or psychiatric illness (acute or chronic) including institution of new medical or surgical treatment or a significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months of screening
* Positive serology for HIV-1 or HIV-2, or HBsAg or HCV antibodies
* Pregnancy or lactation
* Cancer or treatment for cancer, within the previous 3 years, excluding basal cell carcinoma
* Presence of any medical condition that may be associated with impaired immune responsiveness, including diabetes mellitus, per the investigator's discretion
* Presently receiving or history of receiving, during the preceding 3-month period, any medications or other treatments that may adversely affect the immune system

  1. This includes allergy injections, immune globulin, interferon, immunomodulators, cytotoxic drugs, or systemic corticosteroids (oral or injectable; 20 mg/day x 14 days or longer)
  2. Radiation therapy
  3. Intranasal and topical corticosteroids will be allowed
* Receipt or planned administration of a non study vaccine within 14 days prior to vaccination and throughout the study period (30 days for live vaccines) Immunization on an emergency basis with Tetanus Toxoids Adsorbed for adult use (Td or Tdap) or influenza vaccine up to 14 days before or at least 14 days after a dose of study vaccine will be allowed
* History of anaphylactic type reaction to injected vaccines
* History of drug or chemical abuse in the year before the study
* Receipt of any investigational product or nonregistered drug within 30 days prior to vaccination or currently enrolled in any investigational drug study or intends to enroll in such a study within the ensuing study period
* Receipt of blood or blood products 8 weeks prior to vaccination or planned administration during the study period
* Donation of blood or blood products within 8 weeks prior to vaccination or at any time during the study
* Acute disease within 72 hours prior to vaccination

  1. Acute disease is defined as the presence of a moderate or severe illness (as determined by the Investigator through medical history and physical examination) with or without fever (≥38°C; 100.4°F), or an oral temperature of ≥38°C orally
  2. Study vaccine can be administered to persons with a minor illness
* History of immunodeficiency, chronic illness requiring continuous or frequent medical intervention, autoimmune disease, use of immunosuppressive medications, or ongoing therapy with systemic corticosteroids within 3 months prior to any planned vaccine dose. Inhaled and topical steroids are permitted. "Burst" therapy of steroids is permitted except within 2 weeks prior to vaccination.
* Evidence of psychiatric, medical and/or substance abuse problems during the past 6 months that the investigator believes would adversely affect the subject's ability to participate in the trial
* Occupational or other responsibilities that would prevent completion of participation in the trial, including:

  1. US military or reservists who may receive the licensed anthrax vaccine (BioThrax) or served during the Persian Gulf War between January and May, 1991. Such individuals may be enrolled only if they provide their medical records, which can then show proof that they have not received the licensed anthrax vaccine.
  2. Postal and other workers who may be exposed to anthrax or may have to take BioThrax
* Any condition that, in the opinion of the investigator, might interfere with interpretation of data supporting the primary study objectives

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to 3 months

SECONDARY OUTCOMES:
Change from Baseline in antibody titer after three immunizations | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed Army Institute of Research, Clinical Trials Center, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Paolino KM, Regules JA, Moon JE, Ruck RC, Bennett JW, Remich SA, Mills KT, Lin L, Washington CN, Fornillos GA, Lindsey CY, O'Brien KA, Shi M, Mark Jones R, Green BJ, Tottey S, Chichester JA, Streatfield SJ, Yusibov V. Safety and immunogenicity of a plant-derived recombinant protective antigen (rPA)-based vaccine against Bacillus anthracis: A Phase 1 dose-escalation study in healthy adults. Vaccine. 2022 Mar 15;40(12):1864-1871. doi: 10.1016/j.vaccine.2022.01.047. Epub 2022 Feb 10. PMID 35153091